CLINICAL TRIAL: NCT02345161
Title: A Phase III, 24 Week, Randomized, Double Blind, Double Dummy, Parallel Group Study (With an Extension to 52 Weeks in a Subset of Subjects) Comparing the Efficacy, Safety and Tolerability of the Fixed Dose Triple Combination FF/UMEC/VI Administered Once Daily in the Morning Via a Dry Powder Inhaler With Budesonide/Formoterol 400mcg/12mcg Administered Twice-Daily Via a Reservoir Inhaler in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Comparison Study Between the Fixed Dose Triple Combination of Fluticasone Furoate/ Umeclidinium/ Vilanterol Trifenatate (FF/UMEC/VI) With Budesonide/Formoterol in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116853
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Triple Therapy; Formoterol; Respiratory; COPD; Budesonide; Vilanterol; Fluticasone Furoate; Umeclidinium; Lung Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg) (Experimental): Each subject will inhale once from their ELLIPTA DPI and once from the reservoir inhaler in the morning and once from the reservoir inhaler in the evening, for 24 weeks (or 52 weeks for subjects participating in the extension part of the study). Subjects will receive FF/UMEC/VI (100mcg/62.5mcg/25mcg) via the ELLIPTA DPI and placebo via reservoir inhaler.
  Interventions: Drug: Triple FF/UMEC/VI; Drug: Placebo to match FF/UMEC/VI; Drug: Albuterol/salbutamol
- Budesonide/formoterol (400 mcg/12 mcg) (Experimental): Each subject will inhale once from their ELLIPTA DPI and once from the reservoir inhaler in the morning and once from the reservoir inhaler in the evening, for 24 weeks (or 52 weeks for subjects participating in the extension part of the study). Subjects will receive Budesonide/formoterol (400mcg/12mcg) via reservoir inhaler and placebo via the ELLIPTA DPI.
  Interventions: Drug: Budesonide/Formoterol; Drug: Placebo to match Budesonide/Formoterol combination; Drug: Albuterol/salbutamol

INTERVENTIONS:
Drug: Triple FF/UMEC/VI — The combination will be provided as inhalation via an ELLIPTA DPI having 30 doses (2 strips with 30 blisters per strip). It will have 100 mcg of FF (blended with lactose) per blister, 62.5 mcg of UMEC (blended with lactose and magnesium stearate) per blister and 25 mcg of VI (blended with lactose) per blister.
  Arms: FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg)
Drug: Placebo to match FF/UMEC/VI — The placebo (Lactose) will be provided as inhalation via an ELLIPTA DPI having 30 doses (2 strips with 30 blisters per strip).
  Arms: FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg)
Drug: Budesonide/Formoterol — The combination (400 mcg Budesonide/12 mcg Formoterol) will be provided as inhalation via TURBOHALER with 60 doses.
  Arms: Budesonide/formoterol (400 mcg/12 mcg)
Drug: Placebo to match Budesonide/Formoterol combination — The placebo (Lactose) will be provided as inhalation via TURBOHALER with 60 doses.
  Arms: Budesonide/formoterol (400 mcg/12 mcg)
Drug: Albuterol/salbutamol — Albuterol/salbutamol will be available as an inhalation via metered-dose inhaler (MDI) with a spacer and will be issued for reversibility testing at Visit 1 Albuterol/salbutamol MDI or NEBULES™ for as needed (prn) use throughout the study will be provided starting at Visit 1.

SUMMARY:
This is a phase IIIa, randomised, double-blind, double-dummy, parallel group multicenter study evaluating once daily FF/UMEC/VI (100 microgram [mcg]/62.5 mcg/25 mcg) inhalation powder versus twice daily budesonide/formoterol (400 mcg/12 mcg). The primary purpose of this study is to demonstrate improvements in lung function and health status for subjects treated with FF/UMEC/VI compared with budesonide/formoterol for 24 weeks. Once-daily 'closed' triple therapy of a Inhaled Corticosteroid/ Long-acting Muscarinic Receptor Antagonists/ Long Acting Beta-Agonist (ICS/LAMA/LABA) combination FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg) in a single device is being developed with the aim of providing a new treatment option for the management of advanced (GOLD Group D) COPD which will reduce the exacerbation frequency, allow for a reduced burden of polypharmacy, convenience, and increase the potential for improvement in lung function, Health Related Quality of Life (HRQoL) and symptom control over established dual/monotherapies.

Subjects meeting all inclusion/exclusion criteria and who have successfully completed all protocol procedures at the Screening Visit will enter the two-week run-in period. Following the run-in period, eligible subjects will be randomised (1:1) to one of the following double-blind treatment groups: FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg via the ELLIPTA™ dry powder inhaler (DPI) once daily in the morning and placebo via reservoir inhaler twice daily OR Budesonide/formoterol 400 mcg/12 mcg via reservoir inhaler twice daily and placebo via the ELLIPTA DPI once daily in the morning.

The target enrollment is 1800 randomised subjects at approximately 200 study centers globally. The total duration of subject participation will be approximately 27 weeks, consisting of a 2-week run-in period, 24-week treatment period and a 1-week follow-up period. Subjects will run-in on their existing COPD medications for 2 weeks and in addition will be provided with short acting albuterol/salbutamol to be used on an as-needed basis (rescue medication) throughout the study. Subjects will discontinue all existing COPD medications during the randomised treatment period but may continue their study supplied rescue albuterol/salbutamol. A sub-set of approximately 400 subjects will remain on blinded study treatment for up to a total of 52 weeks to provide additional long term safety data.

ELLIPTA and NUBULES are a trade marks of the GlaxoSmithKline Group of Companies. Other company or product names mentioned herein may be the property of their respective owners

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: A signed and dated written informed consent prior to study participation.
* Type of subject: Outpatient.
* Age: Subjects 40 years of age or older at Screening (Visit 1).
* Gender: Male or female subjects. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, >45 years, in the absence of hormone replacement therapy. OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to safety follow-up contact): Abstinence, Oral Contraceptive, either combined or progestogen alone, Injectable progestogen, Implants of levonorgestrel, Estrogenic vaginal ring, Percutaneous contraceptive patches, Intrauterine device (IUD) or intrauterine system (IUS), Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records.; Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* COPD Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >10 pack-years at Screening (Visit 1) [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Note: Pipe and/or cigar use cannot be used to calculate pack-year history.
* Severity of COPD symptoms: A score of >=10 on the COPD Assessment Test (CAT) at Screening (Visit 1).
* Severity of Disease: Subjects must demonstrate at Screening: <a post-bronchodilator FEV1 <50% predicted normal OR a post-bronchodilator FEV1 <80% predicted normal and a documented history of >=2 moderate exacerbations or one severe (hospitalized) exacerbation in the previous 12 months. Subjects must also have a measured post albuterol/salbutamol FEV1/FVC ratio of <0.70 at screening. Note: Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations. Note: A documented history of a COPD exacerbation (e.g., medical record verification) is a medical record of worsening COPD symptoms that required systemic/oral corticosteroids and/or antibiotics (for a moderate exacerbation) or hospitalization (for a severe exacerbation). Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnoea, sputum volume, or sputum purulence (colour). Subject verbal reports are not acceptable.
* Existing COPD maintenance treatment: Subject must be receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening. Note: Subjects receiving only as required (PRN) COPD medications are not eligible.
* Liver function tests: alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase <=1.5xULN; bilirubin <=1.5xULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD). Alpha1-antitrypsin deficiency: Subjects with alpha1-antitrypsin deficiency as the underlying cause of COPD.
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening.
* Risk Factors for Pneumonia: immune suppression (e.g. Human immunodeficiency virus [HIV], Lupus) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis). Subjects at potentially high risk (e.g. very low Body mass index [BMI], severely malnourished, or very low FEV1) will only be included at the discretion of the investigator.
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable). In addition, any subject that experiences pneumonia and/or moderate or severe COPD exacerbation during the run-in period will be excluded.
* Respiratory tract infection that has not resolved at least 7 days prior to Screening.
* Abnormal Chest X-ray (CXR): Chest X-ray (posteroanterior and lateral) reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on CXR (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a CXR at Screening Visit 1) (or historical radiograph or Computed Tomography [CT] scan obtained within 3 months prior to screening) that will be over-read by a central vendor. Note: Subjects who have experienced pneumonia and/or moderate or severe COPD exacerbation within 3 months of screening must provide a post pneumonia/exacerbation CXR to be over-read by the central vendor or have a CXR conducted at Screening. For sites in Germany: If a chest x-ray (or CT scan) within 3 months prior to Screening (Visit 1) is not available, approval to conduct a diagnostic CXR will need to be obtained from the Federal Office for Radiation Protection (BfS).
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study. For subjects taking part in the physical activity monitor subset: Orthopaedic, neurological or other complaints that significantly impair normal biomechanical movement patterns and limit the ability to walk/cycle, as judged by the Investigator.
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria.
* Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure
* Abnormal and clinically significant 12-Lead Electrocardiogram (ECG) finding: Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Principal Investigator (PI) will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: Atrial fibrillation (AF) with rapid ventricular rate >120 Beats Per Minute (BPM); sustained or non-sustained ventricular tachycardia (VT); Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 milliseconds (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.
* Contraindications: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the Investigator, contraindicates study participation.
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment.
* Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3litres/minute (L/min) (Oxygen use <=3L/min flow is not exclusionary.)
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit.
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Affiliation with investigator site: study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Medication prior to screening: No use of the following medications within the following time intervals prior to Screening or during the study. Long term antibiotic therapy: Subjects receiving antibiotics for long term therapy are not eligible for the study (Antibiotics are allowed for the short term treatment of an exacerbation or for short term treatment of other acute infections); Systemic, Oral, parenteral corticosteroids: 30 days (Except during the study oral/systemic corticosteroids may be used to treat COPD exacerbations/pneumonia). Intra-articular injections are allowed. Any other investigational drug: 30 days or 5 half lives whichever is longer.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1811 (Actual)
Dates: Start 2015-01-23; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (121):
- Bulgaria (7):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Lovech
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Vidin
- China (7):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Wuxi
- Czechia (9):
  - GSK Investigational Site, Boskovice
  - GSK Investigational Site, Brandýs nad Labem
  - GSK Investigational Site, Cvikov
  - GSK Investigational Site, Karlovy Vary
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
- Estonia (5):
  - GSK Investigational Site, Haapsalu
  - GSK Investigational Site, Kohtla-Järve
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (15):
  - GSK Investigational Site, Elsterwerda, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Rethymnon, Crete
  - GSK Investigational Site, Thessaloniki
- Hungary (8):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Hatvan
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szikszó
  - GSK Investigational Site, Törökbálint
- Italy (7):
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Varese, Lombardy
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Pisa, Tuscany
- Mexico (11):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Puebla, Pue, Puebla
  - GSK Investigational Site, Cuautitlán Izcalli, State of Mexico
  - GSK Investigational Site, Tlanepantla, State of Mexico
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
  - GSK Investigational Site, Oaxaca City
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Słupsk
- Romania (7):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (16):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Sestroretsk
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Slovakia (5):
  - GSK Investigational Site, Bojnice
  - GSK Investigational Site, Levice
  - GSK Investigational Site, Liptovský Hrádok
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Prešov
- South Korea (4):
  - GSK Investigational Site, Chuncheon
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju-si, Jeollabuk-Do
  - GSK Investigational Site, Seoul
- Ukraine (9):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lipson DA, Birk R, Brealey N, Zhu CQ. 24-Hour Serial Spirometric Assessment of Once-Daily Fluticasone Furoate/Umeclidinium/Vilanterol Versus Twice-Daily Budesonide/Formoterol in Patients with COPD: Analysis of the FULFIL Study. Adv Ther. 2020 Dec;37(12):4894-4909. doi: 10.1007/s12325-020-01496-7. Epub 2020 Oct 3. PMID 33011864
- [Derived] Schroeder M, Benjamin N, Atienza L, Biswas C, Martin A, Whalen JD, Izquierdo Alonso JL, Riesco Miranda JA, Soler-Cataluna JJ, Huerta A, Ismaila AS. Cost-Effectiveness Analysis of a Once-Daily Single-Inhaler Triple Therapy for Patients with Chronic Obstructive Pulmonary Disease (COPD) Using the FULFIL Trial: A Spanish Perspective. Int J Chron Obstruct Pulmon Dis. 2020 Jul 10;15:1621-1632. doi: 10.2147/COPD.S240556. eCollection 2020. PMID 32764908
- [Derived] Mehta R, Farrell C, Hayes S, Birk R, Okour M, Lipson DA. Population Pharmacokinetic Analysis of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2020 Jan;59(1):67-79. doi: 10.1007/s40262-019-00794-w. PMID 31321713
- [Derived] Naya I, Compton C, Ismaila AS, Birk R, Brealey N, Tabberer M, Zhu CQ, Lipson DA, Criner G. Preventing clinically important deterioration with single-inhaler triple therapy in COPD. ERJ Open Res. 2018 Oct 3;4(4):00047-2018. doi: 10.1183/23120541.00047-2018. eCollection 2018 Oct. PMID 30302335
- [Derived] Tabberer M, Lomas DA, Birk R, Brealey N, Zhu CQ, Pascoe S, Locantore N, Lipson DA. Once-Daily Triple Therapy in Patients with COPD: Patient-Reported Symptoms and Quality of Life. Adv Ther. 2018 Jan;35(1):56-71. doi: 10.1007/s12325-017-0650-4. Epub 2018 Jan 8. PMID 29313286
- [Derived] Ismaila AS, Birk R, Shah D, Zhang S, Brealey N, Risebrough NA, Tabberer M, Zhu CQ, Lipson DA. Once-Daily Triple Therapy in Patients with Advanced COPD: Healthcare Resource Utilization Data and Associated Costs from the FULFIL Trial. Adv Ther. 2017 Sep;34(9):2163-2172. doi: 10.1007/s12325-017-0604-x. Epub 2017 Sep 5. PMID 28875459
- [Derived] Lipson DA, Barnacle H, Birk R, Brealey N, Locantore N, Lomas DA, Ludwig-Sengpiel A, Mohindra R, Tabberer M, Zhu CQ, Pascoe SJ. FULFIL Trial: Once-Daily Triple Therapy for Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Aug 15;196(4):438-446. doi: 10.1164/rccm.201703-0449OC. PMID 28375647
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116853 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase IIIa, randomized, double-blind, double-dummy, parallel group multicenter study to evaluate once daily fluticasone furoate (FF)/umeclidinium (UMEC)/vilanterol (VI; 100 micrograms [µg]/62.5 µg/25 µg) inhalation versus twice daily budesonide/formoterol (400 µg/12 µg) in participants with chronic obstructive pulmonary disease.
Pre-assignment Details: A total of 2121 participants were screened in this study and 1811 were randomized following 2-week run-in. Of those, 1 participant was randomized in error and did not receive randomized treatment. This was followed by a 24-week treatment and 1-week follow-up periods. A sub-set of 430 participants continued in a blinded study treatment for 52 weeks.
Groups:
- FF/UMEC/VI 100/62.5/25 µg: Participants received FF/UMEC/VI 100/62.5/25 µg via the ELLIPTA dry powder inhaler (DPI) once daily in the morning and placebo via the Turbuhaler twice daily (BID) for 24 weeks in the treatment period and 52 weeks for participants in the extension part of the study.
- BUD/FOR 400/12 µg: Participants received BUD/FOR 400/12 µg via the Turbuhaler BID and placebo via the ELLIPTA once daily in the morning for 24 weeks in the treatment period and 52 weeks for participants in the extension part of the study.
Period: Overall Study
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Started | 911 | 899
Completed | 866 | 842
Not Completed | 45 | 57
Not completed — Withdrawal by Subject | 25 | 33
Not completed — Adverse Event | 16 | 19
Not completed — Physician Decision | 4 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg | Total
Number analyzed (Participants) | 911 | 899 | 1810
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.56) | 63.7 (8.71) | 63.9 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 236 | 469
  Male | 678 | 663 | 1341
Race/Ethnicity, Customized [Number; unit: Participants]
  Amrican Indian or Alaskan Native | 16 | 19 | 35
  Asian-East Asian Heritage | 55 | 49 | 104
  Asian-South East Asian Heritag | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White-Arabic/North African Heritage | 5 | 8 | 13
  White-White/Caucasina/Euorpean Heritage | 771 | 759 | 1530
  Mixed Race | 63 | 62 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 24
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 at Week 24 was defined as the FEV1 values obtained prior to morning dose of the study treatment. Baseline was defined as the value obtained predose (0 minutes) on Day 1. Change from Baseline was calculated as the pre-dose measurement at Week 24 minus the Baseline value. The analysis was performed using a mixed model repeated measures (MMRM) method including covariates of treatment group, smoking status (screening), geographical region, visit, baseline, baseline by visit and treatment by visit interactions. ITT Population comprised of all randomized subjects excluding those who were randomized in error. Only participants with analyzable data at the given time point were analyzed.
Time Frame: Baseline to Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 836 | 781
Liters (L) | 0.142 (0.0083) | -0.029 (0.0085)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; Adjusted LS mean difference = 0.171, 95% CI 2-sided [0.148 to 0.194], Standard Error of Mean 0.0118

2. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) at Week 52
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 at Week 52 was defined as the FEV1 values obtained prior to morning dose of the study treatment. Baseline was defined as the value obtained predose (0 minutes) on Day 1. Change from Baseline was calculated as the pre-dose measurement at Week 24 minus the Baseline value. The analysis was performed using a mixed model repeated measures (MMRM) method including covariates of treatment group, smoking status (screening), geographical region, visit, baseline, baseline by visit and treatment by visit interactions. Extension Population: all participants in the ITT Population who were enrolled into the subset of participants with extension to 52 weeks.
Time Frame: Baseline to Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 183 | 171
Liters (L) | 0.126 (0.0170) | -0.053 (0.0172)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; Adjusted LS mean difference = 0.179, 95% CI 2-sided [0.131 to 0.226], Standard Error of Mean 0.0242

3. Primary Outcome: Change From Baseline in St George's Respiratory Questionnaire-Chronic Obstructive Pulmonary Disease (COPD; SGRQ) Total Score for COPD Participants at Week 24
Description: The SGRQ-C is a disease-specific questionnaire designed to measure the impact of respiratory disease and its treatment on a COPD participant's health-related quality of life (HRQoL). SGRQ-C total score was converted to SGRQ total score (ranging from 0-100) according to manual. In addition to an overall summary (total) score, scores for the individual domains of Symptoms, Activity, and Impacts (each ranging from 0-100) are produced. A decrease in score indicated improvement in quality of life. The minimum clinically important difference (MCID) for this instrument is a 4-point improvement (decrease from Baseline). Baseline was defined as the value obtained predose on Day 1. Change from Baseline was calculated as total score at Week 24 minus the Baseline value. The analysis for SGRQ total score was performed using a MMRM method including covariates of treatment group, smoking status (screening), geographical region, visit, baseline, baseline by visit and treatment by visit interactions
Time Frame: Baseline to Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 846 | 791
Scores on a scale | -6.6 (0.45) | -4.3 (0.46)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; Adjusted LS mean difference = -2.2, 95% CI 2-sided [-3.5 to -1.0], Standard Error of Mean 0.64

4. Primary Outcome: Change From Baseline in St George's Respiratory Questionnaire-COPD; SGRQ Total Score for COPD Participants at Week 52
Description: The SGRQ-C is a disease-specific questionnaire designed to measure the impact of respiratory disease and its treatment on a COPD participant's health-related quality of life (HRQoL). SGRQ-C total score was converted to SGRQ total score (ranging from 0-100) according to manual. In addition to an overall summary (total) score, scores for the individual domains of Symptoms, Activity, and Impacts (each ranging from 0-100) are produced. A decrease in score indicated improvement in quality of life. The minimum clinically important difference (MCID) for this instrument is a 4-point improvement (decrease from Baseline). Baseline was defined as the value obtained predose on Day 1. Change from Baseline was calculated as total score at Week 52 minus the Baseline value. The analysis for SGRQ total score was performed using a MMRM method including covariates of treatment group, smoking status (screening), geographical region, visit, baseline, baseline by visit and treatment by visit interactions.
Time Frame: Baseline to Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 182 | 174
Scores on a scale | -4.6 (1.01) | -1.9 (1.03)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.065, Mixed Model Repeated Measures; Adjusted LS mean difference = -2.7, 95% CI 2-sided [-5.5 to 0.2], Standard Error of Mean 1.44

5. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score Expressed as Least Square Mean at Week 24
Description: The TDI measures change in the participant's dyspnoea from Baseline. The scores in both indexes depend on ratings for three different categories: functional impairment; magnitude of task; and magnitude of effort. Each of these scales had a possible score ranging from -6 (major deterioration) to +6 (major improvement). TDI focal score was calculated as the sum of the three individual scores and then divided by 2 (so the range of the TDI focal score is -9 to +9). TDI was measured at Week 4 and Week 24. Analysis performed using a repeated measures model with covariates of treatment group, smoking status (screening), geographical region, visit, BDI focal score, BDI focal score by visit and treatment by visit interactions.
Time Frame: Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- FF/UMEC/VI 100/62.5/25 µg: Participants received FF/UMEC/VI 100/62.5/25 µg via the ELLIPTA DPI once daily in the morning and placebo via the Turbuhaler BID for 24 weeks in the treatment period and 52 weeks for participants in the extension part of the study.
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 839 | 788
Scores on a scale | 2.29 (0.096) | 1.72 (0.099)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed effect repeated measures model; LS Mean difference = 0.57, 95% CI 2-sided [0.30 to 0.84], Standard Error of Mean 0.138

6. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score Expressed as Least Square Mean at Week 52
Description: The TDI measures change in the participant's dyspnoea from Baseline. The scores in both indexes depend on ratings for three different categories: functional impairment; magnitude of task; and magnitude of effort. Each of these scales had a possible score ranging from -6 (major deterioration) to +6 (major improvement). TDI focal score was calculated as the sum of the three individual scores and then divided by 2 (so the range of the TDI focal score is -9 to +9). TDI was measured at Weeks 4, 24 and 52. Analysis performed using a repeated measures model with covariates of treatment group, smoking status (screening), geographical region, visit, BDI focal score, BDI focal score by visit and treatment by visit interactions
Time Frame: Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 182 | 174
Scores on a scale | 1.74 (0.221) | 1.39 (0.226)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.279, Mixed effect repeated measures model; LS Mean difference = 0.34, 95% CI 2-sided [-0.28 to 0.97], Standard Error of Mean 0.317

7. Secondary Outcome: Daily Activity Question Percentage of Days Reporting a Score of 2 up to Week 24
Description: Participants were asked to complete the daily activity question as part of the eDiary, which included the following options: 0: fewer activities, 1: no affect on my activities, and 2: more activities than usual. Daily activity question percentage of days with score of 2 over Weeks 1-24 was analysed using an ANCOVA model with covariates of treatment group, smoking status (screening), geographical region and baseline.
Time Frame: Up to Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg) | Budesonide/Formoterol (400 mcg/12 mcg)
Number analyzed (Participants) | 909 | 894
Percentage of days | 0.0 (0.38) | -0.1 (0.39)
Statistical Analysis 1: Comparison: FF/UMEC/VI (100 mcg/62.5 mcg/25 mcg) vs Budesonide/Formoterol (400 mcg/12 mcg); Test type: Superiority or Other; p = 0.817, ANCOVA; LS Mean difference = 0.1, 95% CI 2-sided [-0.9 to 1.1], Standard Error of Mean 0.51

8. Secondary Outcome: Daily Activity Question Percentage of Days Reporting a Score of 2 up to Week 52
Description: Participants were asked to complete the daily activity question as aprt of the eDiary, which included the following options: 0: fewer activities, 1: no affect on my activities, and 2: more activities than usual. Daily activity question percentage of days with score of 2 over Weeks 1-24 was analysed using an ANCOVA model with covariates of treatment group, smoking status (screening), geographical region and baseline.
Time Frame: Up to Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 219
Percentage of days | 0.0 (0.70) | 0.3 (0.69)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.767, ANCOVA; LS Mean difference = -0.3, 95% CI 2-sided [-2.1 to 1.6], Standard Error of Mean 0.95

9. Secondary Outcome: Mean Annual On-treatment Moderate and/or Severe COPD Exacerbations up to Week 24
Description: The mean annual moderate and severe COPD exacerbations during the treatment (trt) period (per participant [par.] per year) was assessed. The event rate for exacerbations was calculated as the number of events x 1000 divided by the total participant exposure during the time-period of interest. An exacerbation of COPD, is defined as the worsening of two or more major symptoms (dyspnea, sputum volume, sputum purulence [color]) for at least two consecutive days; or the worsening of any one major symptom together with any one of the minor symptoms (sore throat, cold, fever without other cause, increased cough, increased wheeze) for at least two consecutive days. Analysis performed using a generalised linear model assuming a negative binomial distribution and covariates of treatment group, exacerbation history (0, 1, >=2 moderate/severe), smoking status (screening), geographical region and post-bronchodilator percent predicted FEV1 (day 1).
Time Frame: Up to Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 907 | 892
Exacerbations per participant per year | 0.22 [0.18 to 0.28] | 0.34 [0.28 to 0.42]
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.002, Generalized linear modeL; Generalized linear model assuming a negative binomial distribution; Rate ratio = 0.65, 95% CI 2-sided [0.49 to 0.86]

10. Secondary Outcome: Mean Annual On-treatment Moderate and/or Severe COPD Exacerbations up to Week 52
Description: as for outcome 9
Time Frame: Up to Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 219
Exacerbations per participant per year | 0.20 [0.15 to 0.28] | 0.36 [0.28 to 0.47]
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.006, Generalized Linear model; Generalized linear model assuming a negative binomial distribution; Rate ratio = 0.56, 95% CI 2-sided [0.37 to 0.85]

11. Secondary Outcome: Assessment of Respiratory Symptoms by Change From Baseline in 4-weekly Mean Exacerbations of Chronic Pulmonary Disease Tool (EXACT)-RS Scores up to Week 24
Description: The EXACT-PRO is a 14 item instrument designed to capture information on the occurrence, frequency, severity, and duration of exacerbations of disease in participants with COPD. EXACT-RS consists of 11 items from the 14 item EXACT-PRO instrument and has a scoring range of 0-40. Three subscales are used to describe different symptoms; dyspnoea (range 0-17), cough and sputum (range 0-11) and chest symptoms (range 0-12). Baseline was defined as the mean value during the period between Visits 1 and 2. Mean scores were calculated for each four weekly period and change from Baseline was calculated as four weekly score minus the Baseline value. Four weekly intervals were analyzed using a MMRM method with covariates of treatment group, smoking status (screening), geographical region, time period, baseline, baseline by time period and treatment by time period interactions. Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title).
Time Frame: Baseline to Week 24
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Scores on a scale
  Week 1-4, n=870,859: number analyzed (Participants) | 870 | 859
  Week 1-4, n=870,859 | -1.45 (0.106) | -0.50 (0.106)
  Week 5-8, n=851,830: number analyzed (Participants) | 851 | 830
  Week 5-8, n=851,830 | -2.00 (0.129) | -0.77 (0.130)
  Week 9-12, n=841,813: number analyzed (Participants) | 841 | 813
  Week 9-12, n=841,813 | -2.23 (0.141) | -1.05 (0.143)
  Week 13-16, n=831,802: number analyzed (Participants) | 831 | 802
  Week 13-16, n=831,802 | -2.42 (0.150) | -1.09 (0.151)
  Week 17-20, n=828,788: number analyzed (Participants) | 828 | 788
  Week 17-20, n=828,788 | -2.43 (0.156) | -1.02 (0.159)
  Week 21-24, n=825,783: number analyzed (Participants) | 825 | 783
  Week 21-24, n=825,783 | -2.31 (0.157) | -0.96 (0.160)
  Breathlessness score, Week 1-4, n=870,859: number analyzed (Participants) | 870 | 859
  Breathlessness score, Week 1-4, n=870,859 | -0.71 (0.057) | -0.20 (0.057)
  Breathlessness score, Week 5-8, n=851,830: number analyzed (Participants) | 851 | 830
  Breathlessness score, Week 5-8, n=851,830 | -0.95 (0.069) | -0.26 (0.070)
  Breathlessness score, Week 9-12, n=841,813: number analyzed (Participants) | 841 | 813
  Breathlessness score, Week 9-12, n=841,813 | -1.03 (0.076) | -0.34 (0.076)
  Breathlessness score, Week 13-16, n=831, 802: number analyzed (Participants) | 831 | 802
  Breathlessness score, Week 13-16, n=831, 802 | -1.11 (0.080) | -0.36 (0.081)
  Breathlessness score, Week 17-20, n=828,788: number analyzed (Participants) | 828 | 788
  Breathlessness score, Week 17-20, n=828,788 | -1.10 (0.084) | -0.31 (0.085)
  Breathlessness score, Week 21-24, n=825,783: number analyzed (Participants) | 825 | 783
  Breathlessness score, Week 21-24, n=825,783 | -1.07 (0.085) | -0.30 (0.087)
  Cough, sputum score, Week 1-4, n=870,859: number analyzed (Participants) | 870 | 859
  Cough, sputum score, Week 1-4, n=870,859 | -0.41 (0.031) | -0.24 (0.031)
  Cough, sputum score, Week 5-8, n=851,830: number analyzed (Participants) | 851 | 830
  Cough, sputum score, Week 5-8, n=851,830 | -0.59 (0.037) | -0.39 (0.038)
  Cough, sputum score, Week 9-12, n=841,813: number analyzed (Participants) | 841 | 813
  Cough, sputum score, Week 9-12, n=841,813 | -0.67 (0.041) | -0.50 (0.041)
  Cough, sputum score, Week 13-16, n=831,802: number analyzed (Participants) | 831 | 802
  Cough, sputum score, Week 13-16, n=831,802 | -0.74 (0.043) | -0.53 (0.043)
  Cough, sputum score, Week 17-20, n=828,788: number analyzed (Participants) | 828 | 788
  Cough, sputum score, Week 17-20, n=828,788 | -0.77 (0.045) | -0.53 (0.045)
  Cough, sputum score, Week 21-24, n=825,783: number analyzed (Participants) | 825 | 783
  Cough, sputum score, Week 21-24, n=825,783 | -0.72 (0.046) | -0.50 (0.046)
  Chest score, Week 1-4, n=870,859: number analyzed (Participants) | 870 | 859
  Chest score, Week 1-4, n=870,859 | -0.33 (0.034) | -0.06 (0.035)
  Chest score, Week 5-8, n=851,830: number analyzed (Participants) | 851 | 830
  Chest score, Week 5-8, n=851,830 | -0.46 (0.042) | -0.12 (0.043)
  Chest score, Week 9-12, n=841,813: number analyzed (Participants) | 841 | 813
  Chest score, Week 9-12, n=841,813 | -0.54 (0.046) | -0.20 (0.047)
  Chest score, Week 13-16, n=831,802: number analyzed (Participants) | 831 | 802
  Chest score, Week 13-16, n=831,802 | -0.58 (0.048) | -0.20 (0.048)
  Chest score, Week 17-20, n=828,788: number analyzed (Participants) | 828 | 788
  Chest score, Week 17-20, n=828,788 | -0.57 (0.050) | -0.17 (0.050)
  Chest score, Week 21-24, n=825,783: number analyzed (Participants) | 825 | 783
  Chest score, Week 21-24, n=825,783 | -0.53 (0.050) | -0.17 (0.051)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.95, 95% CI 2-sided [-1.25 to -0.66], Standard Error of Mean 0.150 — EXACT-RS Scores, Week 1-4
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -1.23, 95% CI 2-sided [-1.59 to -0.87], Standard Error of Mean 0.183 — EXACT-RS Scores, Week 5-8
Statistical Analysis 3: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -1.18, 95% CI 2-sided [-1.57 to -0.78], Standard Error of Mean 0.201 — EXACT-RS Scores, Week 9-12
Statistical Analysis 4: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -1.33, 95% CI 2-sided [-1.75 to -0.91], Standard Error of Mean 0.213 — EXACT-RS Scores, Week 13-16
Statistical Analysis 5: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -1.41, 95% CI 2-sided [-1.85 to -0.97], Standard Error of Mean 0.223 — EXACT-RS Scores, Week 17-20
Statistical Analysis 6: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; Mixed Model Repeated Measures = -1.35, 95% CI 2-sided [-1.79 to -0.91], Standard Error of Mean 0.224 — EXACT-RS Scores, Week 21-24
Statistical Analysis 7: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.52, 95% CI 2-sided [-0.67 to -0.36], Standard Error of Mean 0.080 — Breathlessness EXACT-RS Score, Week 1-4
Statistical Analysis 8: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.69, 95% CI 2-sided [-0.88 to -0.50], Standard Error of Mean 0.098 — Breathlessness EXACT-RS Score, Week 5-8
Statistical Analysis 9: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.69, 95% CI 2-sided [-0.90 to -0.48], Standard Error of Mean 0.108 — Breathlessness EXACT-RS Score, Week 9-12
Statistical Analysis 10: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.75, 95% CI 2-sided [-0.97 to -0.52], Standard Error of Mean 0.115 — Breathlessness EXACT-RS Score, Week 13-16
Statistical Analysis 11: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.79, 95% CI 2-sided [-1.03 to -0.56], Standard Error of Mean 0.120 — Breathlessness EXACT-RS Score, Week 17-20
Statistical Analysis 12: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.77, 95% CI 2-sided [-1.01 to -0.54], Standard Error of Mean 0.122 — Breathlessness EXACT-RS Score, Week 21-24
Statistical Analysis 13: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.17, 95% CI 2-sided [-0.26 to -0.09], Standard Error of Mean 0.044 — Cough and sputum EXACT-RS Score, Week 1-4
Statistical Analysis 14: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.20, 95% CI 2-sided [-0.31 to -0.10], Standard Error of Mean 0.053 — Cough and sputum EXACT-RS Score, Week 5-8
Statistical Analysis 15: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures; LS Mean difference = -0.17, 95% CI 2-sided [-0.28 to -0.05], Standard Error of Mean 0.058 — Cough and sputum EXACT-RS Score, Week 9-12
Statistical Analysis 16: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.22, 95% CI 2-sided [-0.34 to -0.10], Standard Error of Mean 0.061 — Cough and sputum EXACT-RS Score, Week 13-16
Statistical Analysis 17: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.24, 95% CI 2-sided [-0.36 to -0.11], Standard Error of Mean 0.064 — Cough and sputum EXACT-RS Score, Week 17-20
Statistical Analysis 18: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.23, 95% CI 2-sided [-0.35 to -0.10], Standard Error of Mean 0.065 — Cough and sputum EXACT-RS Score, Week 21-24
Statistical Analysis 19: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.27, 95% CI 2-sided [-0.37 to -0.18], Standard Error of Mean 0.049 — Chest EXACT-RS Scores, Week 1-4
Statistical Analysis 20: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.34, 95% CI 2-sided [-0.46 to -0.23], Standard Error of Mean 0.060 — Chest EXACT-RS Scores, Week 5-8
Statistical Analysis 21: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.34, 95% CI 2-sided [-0.47 to -0.21], Standard Error of Mean 0.066 — Chest EXACT-RS Scores, Week 9-12
Statistical Analysis 22: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.38, 95% CI 2-sided [-0.51 to -0.25], Standard Error of Mean 0.068 — Chest EXACT-RS Scores, Week 13-16
Statistical Analysis 23: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.40, 95% CI 2-sided [-0.53 to -0.26], Standard Error of Mean 0.071 — Chest EXACT-RS Scores, Week 17-20
Statistical Analysis 24: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.36, 95% CI 2-sided [-0.50 to -0.22], Standard Error of Mean 0.072 — Chest EXACT-RS Scores, Week 21-24

12. Secondary Outcome: Assessment of Respiratory Symptoms by Change From Baseline in 4-weekly Mean EXACT-RS Scores up to Week 52
Description: as for outcome 11
Time Frame: Baseline to Week 52
Population: Extension Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Scores on a scale
  Week 1-4, n=205, 213: number analyzed (Participants) | 205 | 213
  Week 1-4, n=205, 213 | -1.24 (0.222) | -0.72 (0.218)
  Week 5-8, n=203, 208: number analyzed (Participants) | 203 | 208
  Week 5-8, n=203, 208 | -1.97 (0.265) | -0.90 (0.260)
  Week 9-12, n=201, 206: number analyzed (Participants) | 201 | 206
  Week 9-12, n=201, 206 | -2.18 (0.298) | -1.21 (0.294)
  Week 13-16, n=201, 204: number analyzed (Participants) | 201 | 204
  Week 13-16, n=201, 204 | -2.53 (0.317) | -1.52 (0.313)
  Week 17-20, n=201, 199: number analyzed (Participants) | 201 | 199
  Week 17-20, n=201, 199 | -2.64 (0.342) | -1.53 (0.338)
  Week 21-24, n=202, 197: number analyzed (Participants) | 202 | 197
  Week 21-24, n=202, 197 | -2.63 (0.341) | -1.52 (0.338)
  Week 25-28, n=194, 186: number analyzed (Participants) | 194 | 186
  Week 25-28, n=194, 186 | -2.48 (0.349) | -1.16 (0.347)
  Week 29-32, n=192, 181: number analyzed (Participants) | 192 | 181
  Week 29-32, n=192, 181 | -2.33 (0.350) | -0.90 (0.349)
  Week 33-36, n=187, 180: number analyzed (Participants) | 187 | 180
  Week 33-36, n=187, 180 | -2.12 (0.367) | -0.62 (0.366)
  Week 37-40, n=185, 177: number analyzed (Participants) | 185 | 177
  Week 37-40, n=185, 177 | -2.34 (0.359) | -1.11 (0.358)
  Week 41-44, n=180, 174: number analyzed (Participants) | 180 | 174
  Week 41-44, n=180, 174 | -2.30 (0.363) | -0.81 (0.362)
  Week 45-48, n=180, 173: number analyzed (Participants) | 180 | 173
  Week 45-48, n=180, 173 | -2.17 (0.371) | -0.64 (0.371)
  EXACT-RS Scores, Week 49-52, n=179, 171: number analyzed (Participants) | 179 | 171
  EXACT-RS Scores, Week 49-52, n=179, 171 | -2.03 (0.370) | -0.61 (0.370)
  Breathlessness scores, Week 1-4, n=205, 213: number analyzed (Participants) | 205 | 213
  Breathlessness scores, Week 1-4, n=205, 213 | -0.64 (0.120) | -0.31 (0.118)
  Breathlessness scores, Week 5-8, n=203, 208: number analyzed (Participants) | 203 | 208
  Breathlessness scores, Week 5-8, n=203, 208 | -0.93 (0.147) | -0.32 (0.145)
  Breathlessness scores, Week 9-12, n=201, 206: number analyzed (Participants) | 201 | 206
  Breathlessness scores, Week 9-12, n=201, 206 | -1.05 (0.167) | -0.44 (0.164)
  Breathlessness scores, Week 13-16, n=201, 204: number analyzed (Participants) | 201 | 204
  Breathlessness scores, Week 13-16, n=201, 204 | -1.19 (0.175) | -0.57 (0.173)
  Breathlessness scores, Week 17-20, n=201, 199: number analyzed (Participants) | 201 | 199
  Breathlessness scores, Week 17-20, n=201, 199 | -1.17 (0.189) | -0.50 (0.186)
  Breathlessness scores, Week 21-24, n=202, 197: number analyzed (Participants) | 202 | 197
  Breathlessness scores, Week 21-24, n=202, 197 | -1.13 (0.190) | -0.50 (0.188)
  Breathlessness scores, Week 25-28, n=194, 186: number analyzed (Participants) | 194 | 186
  Breathlessness scores, Week 25-28, n=194, 186 | -1.14 (0.195) | -0.38 (0.194)
  Breathlessness scores, Week 29-32, n=192, 181: number analyzed (Participants) | 192 | 181
  Breathlessness scores, Week 29-32, n=192, 181 | -1.11 (0.196) | -0.26 (0.194)
  Breathlessness scores, Week 33-36, n=187, 180: number analyzed (Participants) | 187 | 180
  Breathlessness scores, Week 33-36, n=187, 180 | -1.08 (0.204) | -0.14 (0.203)
  Breathlessness scores, Week 37-40, n=185, 177: number analyzed (Participants) | 185 | 177
  Breathlessness scores, Week 37-40, n=185, 177 | -1.13 (0.203) | -0.37 (0.202)
  Breathlessness scores, Week 41-44, n=180, 174: number analyzed (Participants) | 180 | 174
  Breathlessness scores, Week 41-44, n=180, 174 | -1.06 (0.208) | -0.24 (0.208)
  Breathlessness scores, Week 45-48, n=180, 173: number analyzed (Participants) | 180 | 173
  Breathlessness scores, Week 45-48, n=180, 173 | -0.97 (0.211) | -0.11 (0.211)
  Breathlessness scores, Week 49-52, n=179, 171: number analyzed (Participants) | 179 | 171
  Breathlessness scores, Week 49-52, n=179, 171 | -0.96 (0.207) | -0.08 (0.207)
  Cough and sputum scores, Week 1-4, n=205, 213: number analyzed (Participants) | 205 | 213
  Cough and sputum scores, Week 1-4, n=205, 213 | -0.34 (0.065) | -0.32 (0.064)
  Cough and sputum scores, Week 5-8, n=203, 208: number analyzed (Participants) | 203 | 208
  Cough and sputum scores, Week 5-8, n=203, 208 | -0.59 (0.076) | -0.44 (0.074)
  Cough and sputum scores, Week 9-12, n=201, 206: number analyzed (Participants) | 201 | 206
  Cough and sputum scores, Week 9-12, n=201, 206 | -0.63 (0.083) | -0.52 (0.082)
  Cough and sputum scores, Week 13-16, n=201, 204: number analyzed (Participants) | 201 | 204
  Cough and sputum scores, Week 13-16, n=201, 204 | -0.73 (0.088) | -0.62 (0.087)
  Cough and sputum scores, Week 17-20, n=201, 199: number analyzed (Participants) | 201 | 199
  Cough and sputum scores, Week 17-20, n=201, 199 | -0.83 (0.095) | -0.73 (0.094)
  Cough and sputum scores, Week 21-24, n=202, 197: number analyzed (Participants) | 202 | 197
  Cough and sputum scores, Week 21-24, n=202, 197 | -0.83 (0.098) | -0.71 (0.097)
  Cough and sputum scores, Week 25-28, n=194, 186: number analyzed (Participants) | 194 | 186
  Cough and sputum scores, Week 25-28, n=194, 186 | -0.73 (0.097) | -0.57 (0.097)
  Cough and sputum scores, Week 29-32, n=192, 181: number analyzed (Participants) | 192 | 181
  Cough and sputum scores, Week 29-32, n=192, 181 | -0.68 (0.096) | -0.48 (0.096)
  Cough and sputum scores, Week 33-36, n=187, 180: number analyzed (Participants) | 187 | 180
  Cough and sputum scores, Week 33-36, n=187, 180 | -0.56 (0.099) | -0.40 (0.099)
  Cough and sputum scores, Week 37-40, n=185, 177: number analyzed (Participants) | 185 | 177
  Cough and sputum scores, Week 37-40, n=185, 177 | -0.65 (0.097) | -0.54 (0.097)
  Cough and sputum scores, Week 41-44, n=180, 174: number analyzed (Participants) | 180 | 174
  Cough and sputum scores, Week 41-44, n=180, 174 | -0.66 (0.101) | -0.41 (0.102)
  Cough and sputum scores, Week 45-48, n=180, 173: number analyzed (Participants) | 180 | 173
  Cough and sputum scores, Week 45-48, n=180, 173 | -0.66 (0.098) | -0.39 (0.099)
  Cough and sputum scores, Week 49-52, n=179, 171: number analyzed (Participants) | 179 | 171
  Cough and sputum scores, Week 49-52, n=179, 171 | -0.61 (0.100) | -0.44 (0.100)
  Chest scores, Week 1-4, n=205, 213: number analyzed (Participants) | 205 | 213
  Chest scores, Week 1-4, n=205, 213 | -0.27 (0.069) | -0.09 (0.068)
  Chest scores, Week 5-8, n=203, 208: number analyzed (Participants) | 203 | 208
  Chest scores, Week 5-8, n=203, 208 | -0.46 (0.084) | -0.13 (0.082)
  Chest scores, Week 9-12, n=201, 206: number analyzed (Participants) | 201 | 206
  Chest scores, Week 9-12, n=201, 206 | -0.51 (0.093) | -0.24 (0.092)
  Chest scores, Week 13-16, n=201, 204: number analyzed (Participants) | 201 | 204
  Chest scores, Week 13-16, n=201, 204 | -0.61 (0.097) | -0.31 (0.095)
  Chest scores, Week 17-20, n=201, 199: number analyzed (Participants) | 201 | 199
  Chest scores, Week 17-20, n=201, 199 | -0.67 (0.104) | -0.29 (0.103)
  Chest scores, Week 21-24, n=202, 197: number analyzed (Participants) | 202 | 197
  Chest scores, Week 21-24, n=202, 197 | -0.68 (0.102) | -0.30 (0.101)
  Chest scores, Week 25-28, n=194, 186: number analyzed (Participants) | 194 | 186
  Chest scores, Week 25-28, n=194, 186 | -0.63 (0.105) | -0.21 (0.104)
  Chest scores, Week 29-32, n=192, 181: number analyzed (Participants) | 192 | 181
  Chest scores, Week 29-32, n=192, 181 | -0.55 (0.107) | -0.16 (0.107)
  Chest scores, Week 33-36, n=187, 180: number analyzed (Participants) | 187 | 180
  Chest scores, Week 33-36, n=187, 180 | -0.48 (0.111) | -0.08 (0.111)
  Chest scores, Week 37-40, n=185, 177: number analyzed (Participants) | 185 | 177
  Chest scores, Week 37-40, n=185, 177 | -0.57 (0.107) | -0.20 (0.107)
  Chest scores, Week 41-44, n=180, 174: number analyzed (Participants) | 180 | 174
  Chest scores, Week 41-44, n=180, 174 | -0.58 (0.108) | -0.16 (0.108)
  Chest scores, Week 45-48, n=180, 173: number analyzed (Participants) | 180 | 173
  Chest scores, Week 45-48, n=180, 173 | -0.57 (0.113) | -0.13 (0.113)
  Chest scores, Week 49-52, n=179, 171: number analyzed (Participants) | 179 | 171
  Chest scores, Week 49-52, n=179, 171 | -0.49 (0.115) | -0.08 (0.115)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.094, Mixed Model Repeated Measures; LS Mean difference = -0.52, 95% CI 2-sided [-1.13 to 0.09], Standard Error of Mean 0.311 — EXACT-RS Scores, Week 1-4
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures; LS Mean difference = -1.07, 95% CI 2-sided [-1.80 to -0.34], Standard Error of Mean 0.371 — EXACT-RS Scores, Week 5-8
Statistical Analysis 3: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.022, Mixed Model Repeated Measures; LS Mean difference = -0.97, 95% CI 2-sided [-1.79 to -0.14], Standard Error of Mean 0.419 — EXACT-RS Scores, Week 9-12
Statistical Analysis 4: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.024, Mixed Model Repeated Measures; LS Mean difference = -1.01, 95% CI 2-sided [-1.88 to -0.13], Standard Error of Mean 0.445 — EXACT-RS Scores, Week 13-16
Statistical Analysis 5: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.021, Mixed Model Repeated Measures; LS Mean difference = -1.11, 95% CI 2-sided [-2.06 to -0.17], Standard Error of Mean 0.481 — EXACT-RS Scores, Week 17-20
Statistical Analysis 6: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.022, Mixed Model Repeated Measures; LS Mean difference = -1.11, 95% CI 2-sided [-2.05 to -0.16], Standard Error of Mean 0.481 — EXACT-RS Score, Week 21-24
Statistical Analysis 7: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.008, Mixed Model Repeated Measures; LS Mean difference = -1.32, 95% CI 2-sided [-2.29 to -0.35], Standard Error of Mean 0.492 — EXACT-RS Scores, Week 25-28
Statistical Analysis 8: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures; LS Mean difference = -1.43, 95% CI 2-sided [-2.40 to -0.46], Standard Error of Mean 0.494 — EXACT-RS Scores, Week 29-32
Statistical Analysis 9: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.004, Mixed Model Repeated Measures; LS Mean difference = -1.50, 95% CI 2-sided [-2.52 to -0.48], Standard Error of Mean 0.519 — EXACT-RS Scores, Week 33-36
Statistical Analysis 10: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.016, Mixed Model Repeated Measures; LS Mean difference = -1.23, 95% CI 2-sided [-2.22 to -0.23], Standard Error of Mean 0.507 — EXACT-RS Scores, Week 37-40
Statistical Analysis 11: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.04, Mixed Model Repeated Measures; LS Mean difference = -1.49, 95% CI 2-sided [-2.50 to -0.48], Standard Error of Mean 0.513 — EXACT-RS Scores, Week 41-44
Statistical Analysis 12: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures; LS Mean difference = -1.53, 95% CI 2-sided [-2.56 to -0.50], Standard Error of Mean 0.525 — EXACT-RS Scores, Week 45-49
Statistical Analysis 13: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures; LS Mean difference = -1.42, 95% CI 2-sided [-2.45 to -0.39], Standard Error of Mean 0.524 — EXACT-RS Scores, Week 49-52
Statistical Analysis 14: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.051, Mixed Model Repeated Measures; LS Mean difference = -0.33, 95% CI 2-sided [-0.66 to 0.00], Standard Error of Mean 0.169 — Breathlessness EXACT-RS score, Week 1-4
Statistical Analysis 15: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.003, Mixed Model Repeated Measures; LS Mean difference = -0.61, 95% CI 2-sided [-1.02 to -0.20], Standard Error of Mean 0.207 — Breathlessness EXACT-RS score, Week 5-8
Statistical Analysis 16: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.010, Mixed Model Repeated Measures; LS Mean difference = -0.61, 95% CI 2-sided [-1.07 to -0.15], Standard Error of Mean 0.234 — Breathlessness EXACT-RS score, Week 9-12
Statistical Analysis 17: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.013, Mixed Model Repeated Measures; LS Mean difference = -0.62, 95% CI 2-sided [-1.10 to -0.13], Standard Error of Mean 0.247 — Breathlessness EXACT-RS score, Week 13-16
Statistical Analysis 18: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.012, Mixed Model Repeated Measures; LS Mean difference = -0.67, 95% CI 2-sided [-1.19 to -0.15], Standard Error of Mean 0.265 — Breathlessness EXACT-RS score, Week 17-20
Statistical Analysis 19: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.018, Mixed Model Repeated Measures; LS Mean difference = -0.64, 95% CI 2-sided [-1.16 to -0.11], Standard Error of Mean 0.268 — Breathlessness EXACT-RS score, Week 21-24
Statistical Analysis 20: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measures; LS Mean difference = -0.76, 95% CI 2-sided [-1.30 to -0.21], Standard Error of Mean 0.275 — Breathlessness EXACT-RS score, Week 25-28
Statistical Analysis 21: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.002, Mixed Model Repeated Measures; LS Mean difference = -0.85, 95% CI 2-sided [-1.40 to -0.31], Standard Error of Mean 0.276 — Breathlessness EXACT-RS score, Week 29-32
Statistical Analysis 22: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.001, Mixed Model Repeated Measures; LS Mean difference = -0.95, 95% CI 2-sided [-1.51 to -0.38], Standard Error of Mean 0.288 — Breathlessness EXACT-RS score, Week 33-36
Statistical Analysis 23: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.008, Mixed Model Repeated Measures; LS Mean difference = -0.76, 95% CI 2-sided [-1.32 to -0.20], Standard Error of Mean 0.287 — Breathlessness EXACT-RS score, Week 37-40
Statistical Analysis 24: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measures; LS Mean difference = -0.82, 95% CI 2-sided [-1.40 to -0.24], Standard Error of Mean 0.294 — Breathlessness EXACT-RS score, Week 41-44
Statistical Analysis 25: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.004, Breathlessness score, Week 41-44; LS Mean difference = -0.85, 95% CI 2-sided [-1.44 to -0.27], Standard Error of Mean 0.299 — Breathlessness EXACT-RS score, Week 45-48
Statistical Analysis 26: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.003, Mixed Model Repeated Measures; LS Mean difference = -0.87, 95% CI 2-sided [-1.45 to -0.30], Standard Error of Mean 0.294 — Breathlessness EXACT-RS score, Week 49-52EXA
Statistical Analysis 27: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.840, Mixed Model Repeated Measures; LS Mean difference = -0.02, 95% CI 2-sided [-0.20 to 0.16], Standard Error of Mean 0.091 — Cough and sputum EXACT-RS score, Week 1-4
Statistical Analysis 28: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.167, Mixed Model Repeated Measures; LS Mean difference = -0.15, 95% CI 2-sided [-0.36 to -0.06], Standard Error of Mean 0.106 — Cough and sputum EXACT-RS score, Week 5-8
Statistical Analysis 29: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.359, Mixed Model Repeated Measures; LS Mean difference = -0.11, 95% CI 2-sided [-0.34 to 0.12], Standard Error of Mean 0.117 — Cough and sputum EXACT-RS score, Week 9-12
Statistical Analysis 30: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.360, Mixed Model Repeated Measures; LS Mean difference = -0.11, 95% CI 2-sided [-0.36 to 0.13], Standard Error of Mean 0.124 — Cough and sputum EXACT-RS score, Week 13-16
Statistical Analysis 31: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.490, Mixed Model Repeated Measures; LS Mean difference = -0.09, 95% CI 2-sided [-0.36 to 0.17], Standard Error of Mean 0.134 — Cough and sputum EXACT-RS score, Week 17-20
Statistical Analysis 32: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.388, Mixed Model Repeated Measures; LS Mean difference = -0.12, 95% CI 2-sided [-0.39 to 0.15], Standard Error of Mean 0.138 — Cough and sputum EXACT-RS score, Week 21-24
Statistical Analysis 33: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.218, Mixed Model Repeated Measures; LS Mean difference = -0.17, 95% CI 2-sided [-0.44 to 0.10], Standard Error of Mean 0.137 — Cough and sputum EXACT-RS score, Week 25-28
Statistical Analysis 34: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.138, Mixed Model Repeated Measures; LS Mean difference = -0.20, 95% CI 2-sided [-0.47 to 0.07], Standard Error of Mean 0.136 — Cough and sputum EXACT-RS score, Week 29-32
Statistical Analysis 35: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.239, Mixed Model Repeated Measures; LS Mean difference = -0.17, 95% CI 2-sided [-0.44 to 0.11], Standard Error of Mean 0.140 — Cough and sputum EXACT-RS score, Week 33-36
Statistical Analysis 36: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.417, Mixed Model Repeated Measures; LS Mean difference = -0.11, 95% CI 2-sided [-0.38 to 0.16], Standard Error of Mean 0.138 — Cough and sputum EXACT-RS score, Week 37-40
Statistical Analysis 37: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.078, Mixed Model Repeated Measures; LS Mean difference = -0.25, 95% CI 2-sided [-0.54 to 0.03], Standard Error of Mean 0.144 — Cough and sputum EXACT-RS score, Week 41-44
Statistical Analysis 38: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.058, Mixed Model Repeated Measures; LS Mean difference = -0.27, 95% CI 2-sided [-0.54 to 0.01], Standard Error of Mean 0.140 — Cough and sputum EXACT-RS score, Week 45-48
Statistical Analysis 39: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.231, Mixed Model Repeated Measures; LS Mean difference = -0.17, 95% CI 2-sided [-0.45 to 0.11], Standard Error of Mean 0.141 — Cough and sputum EXACT-RS score, Week 49-52
Statistical Analysis 40: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.068, Mixed Model Repeated Measures; LS Mean difference = -0.18, 95% CI 2-sided [-0.37 to 0.01], Standard Error of Mean 0.097 — Chest EXACT-RS score, Week 1-4
Statistical Analysis 41: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measures; LS Mean difference = -0.32, 95% CI 2-sided [-0.56 to -0.09], Standard Error of Mean 0.118 — Chest EXACT-RS score, Week 5-8
Statistical Analysis 42: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.042, Mixed Model Repeated Measures; LS Mean difference = -0.27, 95% CI 2-sided [-0.53 to -0.01], Standard Error of Mean 0.131 — Chest EXACT-RS score, Week 9-12
Statistical Analysis 43: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.027, Mixed Model Repeated Measures; LS Mean difference = -0.30, 95% CI 2-sided [-0.57 to -0.03], Standard Error of Mean 0.136 — Chest EXACT-RS score, Week 13-16
Statistical Analysis 44: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.010, Mixed Model Repeated Measures; LS Mean difference = -0.38, 95% CI 2-sided [-0.67 to -0.09], Standard Error of Mean 0.146 — Chest EXACT-RS score, Week 17-20
Statistical Analysis 45: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.010, Mixed Model Repeated Measures; LS Mean difference = -0.37, 95% CI 2-sided [-0.66 to -0.09], Standard Error of Mean 0.144 — Chest EXACT-RS score, Week 21-24
Statistical Analysis 46: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; Mixed Model Repeated Measures; LS Mean difference = -0.41, 95% CI 2-sided [-0.70 to -0.12], Standard Error of Mean 0.148 — Chest EXACT-RS score, Week 25-28
Statistical Analysis 47: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.011, Mixed Model Repeated Measures; LS Mean difference = -0.39, 95% CI 2-sided [-0.68 to -0.09], Standard Error of Mean 0.152 — Chest EXACT-RS score, Week 29-32
Statistical Analysis 48: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.011, Mixed Model Repeated Measures; LS Mean difference = -0.40, 95% CI 2-sided [-0.71 to -0.09], Standard Error of Mean 0.157 — Chest EXACT-RS score, Week 33-36
Statistical Analysis 49: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.014, Mixed Model Repeated Measures; LS Mean difference = -0.37, 95% CI 2-sided [-0.67 to -0.07], Standard Error of Mean 0.151 — Chest EXACT-RS score, Week 37-40
Statistical Analysis 50: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures; LS Mean difference = -0.42, 95% CI 2-sided [-0.72 to -0.12], Standard Error of Mean 0.153 — Chest EXACT-RS score, Week 41-44
Statistical Analysis 51: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.006, Mixed Model Repeated Measures; LS Mean difference = -0.45, 95% CI 2-sided [-0.76 to -0.13], Standard Error of Mean 0.160 — Chest EXACT-RS score, Week 45-48
Statistical Analysis 52: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.013, Mixed Model Repeated Measures; LS Mean difference = -0.41, 95% CI 2-sided [-0.73 to -0.09], Standard Error of Mean 0.163 — Chest EXACT-RS score, Week 49-52

13. Secondary Outcome: Number of Participants With Any On-treatment Adverse Event (AE) and Serious Adverse Event (SAE) in the Treatment Period
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. These included an exacerbation of a chronic or intermittent pre-existing condition. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; or all events of possible drug-induced liver injury. Abnormal and clinically significant laboratory test results were also recorded as an AE or SAE. COPD exacerbations were an expected disease-related outcome and were not to be recorded as an AE, unless they met the definition of an SAE. Participants were not to be withdrawn from the study due to COPD exacerbations and their evaluation was an efficacy endpoint.
Time Frame: Up to Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Participants
  Any AE | 354 | 339
  Any SAE | 49 | 51

14. Secondary Outcome: Number of Participants With Any On-treatment AE/SAEs in the Extension Part of the Study
Description: as for outcome 13
Time Frame: Up to Week 52
Population: Extension Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Participants
  Any AE | 100 | 122
  Any SAE | 21 | 28

15. Secondary Outcome: Number of Participants With an On-treatment Penumonia Event in the Treatment Period
Description: All suspected pneumonias required confirmation as defined by the presence of new infiltrate(s) on chest x-ray and at least 2 of the following signs and symptoms: Increased cough, Increased sputum purulence (colour) or production, Auscultatory findings of adventitious sounds , Dyspnea or tachypnea, Fever (oral temperature > 37.5 °C), Elevated white blood cells (WBC) (>10,000/millimeter [mm^3] or >15 percent immature forms) or Hypoxemia (hemoglobin/oxygen [HbO2] saturation <88 percent or at least 2 percent lower than Baseline value).
Time Frame: Up to Week 24
Population: ITT Population.
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Participants | 20 | 7

16. Secondary Outcome: Number of Participants With an On-treatment Penumonia Event in the Extension Part of the Study
Description: All suspected pneumonias required confirmation as defined by the presence of new infiltrate(s) on chest x-ray AND at least 2 of the following signs and symptoms: Increased cough, Increased sputum purulence (colour) or production, Auscultatory findings of adventitious sounds , Dyspnea or tachypnea, Fever (oral temperature > 37.5 °C), Elevated WBC (>10,000/mm3 or >15 percent immature forms) orr Hypoxemia (HbO2 saturation <88 percent or at least 2 percent lower than Baseline value).
Time Frame: Up to Week 52
Population: Extension Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Participants | 4 | 4

17. Secondary Outcome: Number of Participants With Any On-treatment Cardiovascular (CV) Events (Including Supraventricular Arrhythmia and Non Fatal Myocardial Infarction) in the Treatment Period
Description: Cardiovascular safety was monitored via AE reporting with categorization and analysis of adverse events of special interest (AESIs) including cardiac arrhythmia, cardiac failure, ischemic heart disease, hypertension, and central nervous system hemorrhages and cerebrovascular conditions. In addition, ECGs and vital signs were measured in all subjects and24-hour Holter monitoring was performed in a predefined subset. Pre-specified MACE analysis was conducted based on adjudicated CV deaths and investigator-reported non-fatal AEs. Number of participants with any of the following MACE events were to be included per the broad and narrow analyses: Broad MACE criteria (ischemic heart disease standardized MedDRA query [SMQ; myocardial infarction SMQ and other ischemic diseases]) and narrow MACE criteria (myocardial infarction [acute myocardial infarction].
Time Frame: Up to Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Participants
  Any MACE, Narrow definition | 4 | 7
  Any MACE, Broad definition | 12 | 11

18. Secondary Outcome: Number of Participants With Any On-treatment CV Events (Including Supraventricular Arrhythmia and Non Fatal Myocardial Infarction) in the Extension Part of the Study
Description: as for outcome 17
Time Frame: Up to Week 52
Population: Extension Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Participants
  Any MACE, Narrow definition | 5 | 2
  Any MACE, Broad definition | 7 | 5

19. Secondary Outcome: Change From Baseline in Heart Rate at Week 24
Description: A single 12-lead electrocardiogram (ECG) and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4 and Week 24 or IP Discontinuation Visit. Change from Baseline in ECG heart rate was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value at Week 24 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). All ECG measurements were made with the participants in a supine position having rested in this position for approximately 5 minutes before each reading.
Time Frame: Baseline and Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (Bpm)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 840 | 787
Beats per minute (Bpm) | -1.1 (11.51) | -1.2 (10.91)

20. Secondary Outcome: Change From Baseline in Heart Rate at Week 52
Description: A single 12-lead ECG and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4, Week 24 and Week 52 or IP Discontinuation Visit. Change from Baseline in ECG heart rate was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value at Week 52 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). All ECG measurements were made with the participants in a supine position having rested in this position for approximately 5 minutes before each reading.
Time Frame: Baseline and Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (Standard Deviation); unit: Bpm
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 181 | 169
Bpm | 0.2 (11.30) | -1.0 (10.77)

21. Secondary Outcome: Change From Baseline in Corrected QT Interval Using Fridericia's Correction (QTcF) and PR Interval at Week 24
Description: A single 12-lead ECG and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4 and Week 24 or IP Discontinuation Visit. Change from Baseline in ECG QTcF and PR interval was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value at Week 24 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). All ECG measurements were made with the participants in a supine position having rested in this position for approximately 5 minutes before each reading.
Time Frame: Baseline and Week 24
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Milliseconds (msec)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Milliseconds (msec)
  QTcF, n=840,787: number analyzed (Participants) | 840 | 787
  QTcF, n=840,787 | 2.5 (0.56) | 0.6 (0.58)
  PR, n=812,766: number analyzed (Participants) | 812 | 766
  PR, n=812,766 | -0.1 (0.54) | 0.5 (0.56)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.023, Mixed Model Repeated Measures; LS mean difference = 1.8, 95% CI 2-sided [0.3 to 3.4], Standard Error of Mean 0.81 — For QTcF
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.471, Mixed Model Repeated Measures; LS mean difference = -0.6, 95% CI 2-sided [-2.1 to 1.0], Standard Error of Mean 0.78 — For PR interval

22. Secondary Outcome: Change From Baseline in QTcF and PR Interval at Week 52
Description: Single 12-lead ECG and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4, Week 24 and Week 52 or IP Discontinuation Visit. Change from Baseline in ECG QTcF and PR interval was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value at Week 52 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title).
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Msec
  QTcF, n=181,169: number analyzed (Participants) | 181 | 169
  QTcF, n=181,169 | 1.4 (1.27) | 2.4 (1.31)
  PR, n=174,160: number analyzed (Participants) | 174 | 160
  PR, n=174,160 | 1.6 (1.09) | 1.4 (1.13)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.564, Mixed Model Repeated Measures; LS mean difference = -1.1, 95% CI 2-sided [-4.7 to 2.5], Standard Error of Mean 1.83 — For QTcF
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.908, Mixed Model Repeated Measures; LS mean difference = 0.2, 95% CI 2-sided [-2.9 to 3.3], Standard Error of Mean 1.57 — For PR interval

23. Secondary Outcome: Change From Baseline in QT Interval Corrected for Heart Rate According to Bazett's Formula (QTcB) at Week 24
Description: A single 12-lead ECG and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4 and Week 24 or IP Discontinuation Visit. Change from Baseline in QTcB was summarized for each post-Baseline assessment up to Week 24. Change from Baseline was calculated as the individual post-Baseline value at Week 24 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). All ECG measurements were made with the participants in a supine position having rested in this position for approximately 5 minutes before each reading.
Time Frame: Baseline and Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (Standard Deviation); unit: Msec
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 840 | 787
Msec | 1.5 (21.00) | -0.7 (20.48)

24. Secondary Outcome: Change From Baseline in QTcB at Week 52
Description: A single 12-lead ECG and rhythm strip were recorded after measurement of vital signs and spirometry. Recordings were made at Screening (Visit 1) and approximately 15-45 minutes after dosing on treatment Week 4, Week 24, and Week 52 or IP Discontinuation Visit. Change from Baseline in QTcB was summarized for each post-Baseline assessment up to Week 52. Change from Baseline was calculated as the individual post-Baseline value at Week 52 minus the Baseline value. Baseline value is defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). All ECG measurements were made with the participants in a supine position having rested in this position for approximately 5 minutes before each reading.
Time Frame: Baseline and Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Mean (Standard Deviation); unit: Msec
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 181 | 169
Msec | 0.9 (21.30) | 2.2 (22.46)

25. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressures (BP) at Week 24
Description: Vital signs were obtained at the Screening Visit and prior to taking the morning dose of study treatment and prior to conducting spirometry at Week 4 and Week 24 or at the Study Treatment Discontinuation Visit. A single set of blood pressure (systolic and diastolic) measurements were collected taken after the participant had rested for 5 minutes in the sitting position. Change from Baseline values for systolic and diastolic BP (SBP and DBP) at Week 24 were summarised and these data were analyzed using MMRM analysis. Baseline was defined as the values from most recent assessment prior to randomization which records both systolic and diastolic BP (generally Screening but could be a test repeat).
Time Frame: Baseline and Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 855 | 805
Millimeter of mercury (mmHg)
  SBP | -1.0 (0.39) | -1.1 (0.40)
  DBP | -0.3 (0.27) | -0.5 (0.27)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.849, Mixed Model Repeated Measures; LS mean difference = 0.1, 95% CI 2-sided [-1.0 to 1.2], Standard Error of Mean 0.56 — Week 24, SBP
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.613, Mixed Model Repeated Measures; LS mean difference = 0.2, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.38 — Week 24, DBP

26. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressures (BP) at Week 52
Description: Vital signs were obtained at the Screening Visit and prior to taking the morning dose of study treatment and prior to conducting spirometry at Week 4, Week 24, and Week 52 or at the Study Treatment Discontinuation Visit. A single set of blood pressure (systolic and diastolic) measurements were taken after the participant had rested for 5 minutes in the sitting position. Change from Baseline values for systolic and diastolic BP (SBP and DBP) at Week 52 were summarised and these data were analyzed using MMRM analysis. Baseline was defined as the values from most recent assessment prior to randomization which records both systolic and diastolic BP (generally Screening but could be a test repeat).
Time Frame: Baseline and Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 184 | 175
mmHg
  SBP | -1.3 (0.83) | 0.3 (0.85)
  DBP | -0.4 (0.52) | 0.4 (0.53)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.183, Mixed Model Repeated Measures; : LS mean difference = -1.6, 95% CI 2-sided [-3.9 to 0.8], Standard Error of Mean 1.19 — Week 52, SBP
Statistical Analysis 2: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.253, Mixed Model Repeated Measures; LS mean difference = -0.9, 95% CI 2-sided [-2.3 to 0.6], Standard Error of Mean 0.75 — Week 52, DBP

27. Secondary Outcome: Number of Participants With Any Abnormal Holter Electrocardiogram (ECG) Finding at Week 24
Description: The 24-hour holter measurements were obtained at Screening and 24 hours prior to Week 24 (Visits 1 and 6). The number of participants with clinically significant change (abnormal) were reported. Holter Monitoring Population: all participants in the ITT Population who had at least one holter monitoring evaluation.
Time Frame: Up to Week 24
Population: Holter Monitoring Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Number; unit: Participants
Groups:
- Overall Study Arm: Participants received FF/UMEC/VI 100/62.5/25 µg via the ELLIPTA DPI once daily in the morning and placebo via the Turbuhaler BID for 24 weeks in the treatment period and 52 weeks for participants in the extension part of the study.
Arm/Group | Overall Study Arm | BUD/FOR 400/12 µg
Number analyzed (Participants) | 212 | 206
Participants | 180 | 165

28. Secondary Outcome: Change From Baseline in Pulse Rate at Week 24
Description: Pulse rate was obtained at the Screening Visit and prior to taking the morning dose of study treatment and prior to conducting spirometry at Week 4 and Week 24 or at the Study Treatment Discontinuation. Pulse rate was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from Baseline values for pulse rate at Week 24 were summarised and these data were analyzed using MMRM analysis. Baseline was defined as the values from most recent assessment prior to randomization (generally Screening but could be a test repeat).
Time Frame: Baseline and Week 24
Population: ITT Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Bpm
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 855 | 805
Bpm | -0.5 (0.31) | -0.8 (0.32)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.526, Mixed Model Repeated Measures; LS mean difference = 0.3, 95% CI 2-sided [-0.6 to 1.2], Standard Error of Mean 0.45

29. Secondary Outcome: Change From Baseline in Pulse Rate at Week 52
Description: Pulse rate was obtained at the Screening Visit and prior to taking the morning dose of study treatment and prior to conducting spirometry at Week 4, Week 24, and Week 52 or at the Study Treatment Discontinuation. Pulse rate was measured in a sitting position after the participant was kept at rest for at least 5 minutes. Change from Baseline values for pulse rate at Week 52 were summarized and these data were analyzed using MMRM analysis. Baseline was defined as the values from most recent assessment prior to randomization (generally Screening but could be a test repeat).
Time Frame: Baseline and Week 52
Population: Extension Population; Only participants with analyzable data at the given time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Bpm
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 184 | 175
Bpm | 0.7 (0.67) | -1.9 (0.69)
Statistical Analysis 1: Comparison: FF/UMEC/VI 100/62.5/25 µg vs BUD/FOR 400/12 µg; Test type: Superiority or Other; p = 0.007, Mixed Model Repeated Measures; LS mean difference = 2.6, 95% CI 2-sided [0.7 to 4.5], Standard Error of Mean 0.96

30. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Monocytes, Neutrophils, Leukocytes, Lymphocytes, and Platelets at Week 24
Description: Hematology laboratory assessments included basophils, eosinophils, lymphocytes, monocytes, neutrophils, total neutrophil, leukocytes, and platelets; parameters were measured at Baseline (BL), Week 12 and Week 24. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose value at Week 24. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a repeat test). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter(L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
10^9 cells/Liter(L)
  Week 24, Basophils, n=817,761: number analyzed (Participants) | 817 | 761
  Week 24, Basophils, n=817,761 | -0.001 (0.0217) | -0.001 (0.0204)
  Maximum post BL, Basophils, n=876,853: number analyzed (Participants) | 876 | 853
  Maximum post BL, Basophils, n=876,853 | 0.005 (0.0211) | 0.005 (0.0206)
  Week 24, Eosinophils, n=817, 761: number analyzed (Participants) | 817 | 761
  Week 24, Eosinophils, n=817, 761 | -0.008 (0.1926) | -0.015 (0.1926)
  Maxmium post BL, Eosinophils, n=876,853: number analyzed (Participants) | 876 | 853
  Maxmium post BL, Eosinophils, n=876,853 | 0.034 (0.1941) | 0.019 (0.1952)
  Category title 5. Week 24, Monocytes, n=817,761: number analyzed (Participants) | 817 | 761
  Category title 5. Week 24, Monocytes, n=817,761 | -0.006 (0.1977) | 0.004 (0.2125)
  Maximum post BL, Monocytes, n=876,853: number analyzed (Participants) | 876 | 853
  Maximum post BL, Monocytes, n=876,853 | 0.040 (0.1985) | 0.048 (0.2069)
  Week 24, Neutrophils, n=817,761: number analyzed (Participants) | 817 | 761
  Week 24, Neutrophils, n=817,761 | 0.071 (1.7682) | 0.142 (1.8552)
  Maximum post BL, Neutrophils, n=876,853: number analyzed (Participants) | 876 | 853
  Maximum post BL, Neutrophils, n=876,853 | 0.481 (1.8761) | 0.649 (1.9143)
  Week 24, Leukocytes, n=819,761: number analyzed (Participants) | 819 | 761
  Week 24, Leukocytes, n=819,761 | 0.06 (1.847) | 0.11 (1.915)
  Maximum post BL, Leukocytes, n=877,853: number analyzed (Participants) | 877 | 853
  Maximum post BL, Leukocytes, n=877,853 | 0.52 (1.940) | 0.64 (1.947)
  Week 24, Platelets, n=810,759: number analyzed (Participants) | 810 | 759
  Week 24, Platelets, n=810,759 | -0.7 (43.12) | -0.7 (44.26)
  Maximum post BL, Platelets, n=871,846: number analyzed (Participants) | 871 | 846
  Maximum post BL, Platelets, n=871,846 | 10.8 (42.50) | 10.2 (45.46)
  Week 24, Lymphocytes, n=817,761: number analyzed (Participants) | 817 | 761
  Week 24, Lymphocytes, n=817,761 | 0.002 (0.5311) | -0.023 (0.5669)
  Maximum post BL, Lymphocytes, n=876,853: number analyzed (Participants) | 876 | 853
  Maximum post BL, Lymphocytes, n=876,853 | 0.187 (0.5468) | 0.150 (0.5767)

31. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Monocytes, Neutrophils, Leukocytes, Lymphocytes, and Platelets at Week 52
Description: Hematology laboratory assessments included Basophils, eosinophils, lymphocytes, monocytes,neutrophils, total neutrophil, leukocytes, and platelets; parameters were measured at Baseline (BL), Week 12, Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose value at Week 52. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
10^9 cells/L
  Week 52, Basophils, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Basophils, n=168,166 | 0.002 (0.0203) | 0.003 (0.0241)
  Maximum post BL, Basophils, n=205,212: number analyzed (Participants) | 205 | 212
  Maximum post BL, Basophils, n=205,212 | 0.011 (0.0196) | 0.010 (0.0226)
  Week 52, Eosinophils, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Eosinophils, n=168,166 | 0.002 (0.1819) | -0.011 (0.2567)
  Maximum post BL, Eosinophils, n=205,212: number analyzed (Participants) | 205 | 212
  Maximum post BL, Eosinophils, n=205,212 | 0.074 (0.2460) | 0.057 (0.2884)
  Week 52, Monocytes, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Monocytes, n=168,166 | 0.025 (0.2382) | 0.028 (0.2164)
  Maximum post BL, Monocytes, n=205,212: number analyzed (Participants) | 205 | 212
  Maximum post BL, Monocytes, n=205,212 | 0.075 (0.2359) | 0.072 (0.2123)
  Week 52, Neutrophils, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Neutrophils, n=168,166 | 0.246 (2.1768) | -0.163 (2.3222)
  Maximum post BL, Neutrophils, n=205,212: number analyzed (Participants) | 205 | 212
  Maximum post BL, Neutrophils, n=205,212 | 0.923 (2.1444) | 0.835 (2.1223)
  Week 52, Leukocytes, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Leukocytes, n=168,166 | 0.33 (2.243) | -0.17 (2.387)
  Maximum post BL, Leukocytes, n=205,212: number analyzed (Participants) | 205 | 212
  Maximum post BL, Leukocytes, n=205,212 | 0.97 (2.163) | 0.87 (2.168)
  Week 52, Platelets, n=170,166: number analyzed (Participants) | 170 | 166
  Week 52, Platelets, n=170,166 | -1.8 (39.96) | -2.7 (49.22)
  Maximum post BL, Platelets, n=203,210: number analyzed (Participants) | 203 | 210
  Maximum post BL, Platelets, n=203,210 | 13.6 (40.57) | 13.9 (51.61)
  Week 52, Lymphocytes, n=168,166: number analyzed (Participants) | 168 | 166
  Week 52, Lymphocytes, n=168,166 | 0.060 (0.6850) | -0.027 (0.5714)
  Maximum post BL, Lymphocytes, n=202,212: number analyzed (Participants) | 202 | 212
  Maximum post BL, Lymphocytes, n=202,212 | 0.325 (0.6299) | 0.295 (0.5910)

32. Secondary Outcome: Change From Baseline in Erythrocytes at Week 24
Description: Hematology laboratory assessments included erythrocytes and was measured at Baseline, Week 12 and Week 24. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose value at Week 24. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
10^12 cells/L
  Week 24, n=822,769: number analyzed (Participants) | 822 | 769
  Week 24, n=822,769 | -0.02 (0.292) | -0.04 (0.294)
  Maximum post BL, n=880,857: number analyzed (Participants) | 880 | 857
  Maximum post BL, n=880,857 | 0.06 (0.270) | 0.04 (0.273)

33. Secondary Outcome: Change From Baseline in Erythrocytes at Week 52
Description: Hematology laboratory assessments included erythrocytes and was measured at Baseline, Week 12 and Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated by subtracting the Baseline value from the individual post-dose value at Week 52. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
10^12 cells/L
  Week 52, n=174,170: number analyzed (Participants) | 174 | 170
  Week 52, n=174,170 | 0.02 (0.282) | 0.00 (0.313)
  Maximum post BL, n=206,212: number analyzed (Participants) | 206 | 212
  Maximum post BL, n=206,212 | 0.11 (0.261) | 0.07 (0.289)

34. Secondary Outcome: Change From Baseline in Hemoglobin at Week 24
Description: Blood samples were collected for the measurement of hemoglobin at Baseline, Week 12, and Week 24. Change from Baseline was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Grams per liter (g/L)
  Week 24, n=822,769 | -0.9 (8.17) | -1.0 (8.65)
  Maximum post BL, n=880,857 | 1.5 (7.55) | 1.5 (8.26)

35. Secondary Outcome: Change From Baseline in Hemoglobin at Week 52
Description: Blood samples were collected for the measurement of hemoglobin at Baseline, Week 12, Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated as the post-Baseline value at Week 52 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
g/L
  Week 52, n=174,170: number analyzed (Participants) | 174 | 170
  Week 52, n=174,170 | -2.5 (8.06) | -2.5 (9.82)
  Maximum post BL, n=206,212: number analyzed (Participants) | 206 | 212
  Maximum post BL, n=206,212 | 2.2 (7.67) | 1.9 (8.55)

36. Secondary Outcome: Change From Baseline in Hematocrit at Week 24
Description: Blood samples were collected for the measurement of hematocrit (proportion of red blood cells in blood) at Baseline, Week 12, and Week 24. Change from Baseline was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Fraction of 1
  Week 24, n=822,769: number analyzed (Participants) | 822 | 769
  Week 24, n=822,769 | 0.0024 (0.02627) | 0.0024 (0.02798)
  Maximum post BL, n=880,857: number analyzed (Participants) | 880 | 857
  Maximum post BL, n=880,857 | 0.0115 (0.02533) | 0.0123 (0.02669)

37. Secondary Outcome: Change From Baseline in Hematocrit at Week 52
Description: Blood samples were collected for the measurement of hematocrit (proportion of red blood cells in blood) at Baseline, Week 12, Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as Most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Fraction of 1
  Week 52, n=174,170: number analyzed (Participants) | 174 | 170
  Week 52, n=174,170 | -0.0056 (0.02468) | -0.0056 (0.03170)
  Maximum post BL, n=206,212: number analyzed (Participants) | 206 | 212
  Maximum post BL, n=206,212 | 0.0153 (0.02552) | 0.0149 (0.02793)

38. Secondary Outcome: Change From Baseline in Albumin and Protein at Week 24
Description: Blood samples were collected for the measurement of albumin and protein at Baseline, Week 12 and Week 24. Change from Baseline (BL) was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). The maximum post BL values have been presented. Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
g/L
  Week 24, Albumin, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Albumin, n=839,787 | -0.7 (2.55) | -0.5 (2.41)
  Maximum post BL, Albumin, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Albumin, n=888,866 | 0.1 (2.36) | 0.2 (2.24)
  Week 24, Protein, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Protein, n=839,787 | -0.6 (3.70) | -1.0 (3.64)
  Maximum post BL, Protein, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Protein, n=888,866 | 0.4 (3.42) | 0.1 (3.43)

39. Secondary Outcome: Change From Baseline in Albumin and Protein at Week 52
Description: Blood samples were collected for the measurement of albumin and protein at Baseline, Week 12, Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated as the post-Baseline value at Week 52 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
g/L
  Week 52, Albumin, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Albumin, n=181,174 | -0.8 (2.77) | -0.7 (2.64)
  Maximum post BL,Albumin, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Albumin, n=207,214 | 0.4 (2.45) | 0.2 (2.25)
  Week 52, Protein, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Protein, n=181,174 | -1.1 (4.04) | -1.6 (3.86)
  Maximum post BL, Protein, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Protein, n=207,214 | 0.6 (3.57) | 0.0 (3.30)

40. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Aminotransferase (GGT), Alkaline Phosphatase (ALP), and Creatine Kinase at Week 24
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK, and GGT at Baseline, Week 12 and Week 24. Change from Baseline was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
International units per liter (IU/L)
  Week 24, ALT, n=838,785: number analyzed (Participants) | 838 | 785
  Week 24, ALT, n=838,785 | 1.4 (10.81) | 3.8 (69.15)
  Maximum post BL, ALT, n=887,864: number analyzed (Participants) | 887 | 864
  Maximum post BL, ALT, n=887,864 | 3.0 (11.99) | 5.5 (66.01)
  Week 24, AST, n=835,785: number analyzed (Participants) | 835 | 785
  Week 24, AST, n=835,785 | 1.1 (10.30) | 4.0 (86.63)
  Maximum post BL, AST, n=887,866: number analyzed (Participants) | 887 | 866
  Maximum post BL, AST, n=887,866 | 3.2 (12.61) | 5.6 (82.66)
  Week 24, ALP, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, ALP, n=839,787 | 1.1 (15.42) | -2.8 (12.47)
  Maximum post BL, ALP, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, ALP, n=888,866 | 4.3 (16.46) | 0.8 (11.96)
  Week 24, GGT, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, GGT, n=839,787 | 3.4 (31.65) | 0.5 (21.84)
  Maximum post BL, GGT, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, GGT, n=888,866 | 7.5 (42.66) | 4.7 (27.76)
  Week 24, Creatine Kinase, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Creatine Kinase, n=839,787 | -3.9 (106.48) | -3.4 (191.25)
  Maximum post BL, Creatine Kinase, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Creatine Kinase, n=888,866 | 20.6 (138.17) | 20.6 (185.06)

41. Secondary Outcome: Change From Baseline in ALT, AST, GGT, ALP, and Creatine Kinase at Week 52
Description: Blood samples were collected for the measurement of ALP, ALT, AST, CK, and GGT at Baseline, Week 12, Week 24 and Week 52 for the extension part of the study. Change from Baseline was calculated as the post-Baseline value at Week 52 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
International units per liter (IU/L)
  Week 52, ALT, n=181,173: number analyzed (Participants) | 181 | 173
  Week 52, ALT, n=181,173 | 1.7 (10.64) | 1.3 (12.38)
  Maximum post BL, ALT, n=207,212: number analyzed (Participants) | 207 | 212
  Maximum post BL, ALT, n=207,212 | 5.4 (15.45) | 4.5 (12.84)
  Week 52, AST, n=180,174: number analyzed (Participants) | 180 | 174
  Week 52, AST, n=180,174 | 1.7 (9.72) | 0.8 (11.16)
  Maximum post BL, AST, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, AST, n=207,214 | 5.5 (15.55) | 3.7 (11.65)
  Week 52, ALP, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, ALP, n=181,174 | 1.7 (13.77) | -2.7 (10.83)
  Maximum post BL, ALP, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, ALP, n=207,214 | 6.7 (12.84) | 1.2 (11.73)
  Week 52, GGT, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, GGT, n=181,174 | 0.2 (28.77) | 0.2 (26.86)
  Maximum post BL, GGT, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, GGT, n=207,214 | 7.7 (31.33) | 8.9 (34.98)
  Week 52, Creatine Kinase, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Creatine Kinase, n=181,174 | 6.1 (68.48) | 16.7 (97.17)
  Maximum post BL, Creatine Kinase, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Creatine Kinase, n=207,214 | 39.9 (79.71) | 46.9 (90.78)

42. Secondary Outcome: Change From Baseline in Glucose, Calcium, Carbon Dioxide (CO2), Chloride, Phosphate, Potassium, Sodium, and Urea at Week 24
Description: Blood samples were collected for the measurement of Glucose, calcium, CO2, chloride, phophate, potassium, sodium, and urea at Baseline, Week 12, and Week 24. Change from Baseline was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Millimoles per liter (mmol/L)
  Week 24, Calcium, n=835,785: number analyzed (Participants) | 835 | 785
  Week 24, Calcium, n=835,785 | -0.016 (0.0887) | -0.014 (0.0931)
  Maximum post BL, Calcium, n=887,866: number analyzed (Participants) | 887 | 866
  Maximum post BL, Calcium, n=887,866 | 0.013 (0.0817) | 0.012 (0.0868)
  Week 24, Chloride, n=838,787: number analyzed (Participants) | 838 | 787
  Week 24, Chloride, n=838,787 | -0.4 (2.76) | -0.7 (2.60)
  Maximum post BL, Chloride, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Chloride, n=888,866 | 0.9 (2.53) | 0.6 (2.35)
  Week 24, CO2, n=835,785: number analyzed (Participants) | 835 | 785
  Week 24, CO2, n=835,785 | -0.6 (2.54) | -0.0 (2.61)
  Maximum post BL, CO2, n=835,785: number analyzed (Participants) | 835 | 785
  Maximum post BL, CO2, n=835,785 | 0.0 (2.38) | 0.5 (2.48)
  Week 24, Glucose, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Glucose, n=839,787 | 0.12 (1.433) | -0.00 (1.449)
  Maximum post BL, Glucose, n=887,866: number analyzed (Participants) | 887 | 866
  Maximum post BL, Glucose, n=887,866 | 0.53 (1.506) | 0.37 (1.463)
  Week 24, Potassium, n=834,785: number analyzed (Participants) | 834 | 785
  Week 24, Potassium, n=834,785 | 0.04 (0.457) | -0.03 (0.456)
  Maximum post BL, Potassium, n=887,866: number analyzed (Participants) | 887 | 866
  Maximum post BL, Potassium, n=887,866 | 0.18 (0.428) | 0.13 (0.417)
  Week 24, Phosphate, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Phosphate, n=839,787 | -0.028 (0.2373) | -0.029 (0.2728)
  Maximum post BL, Phosphate, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Phosphate, n=888,866 | 0.039 (0.2310) | 0.043 (0.2576)
  Week 24, Sodium, n=837,787: number analyzed (Participants) | 837 | 787
  Week 24, Sodium, n=837,787 | -0.3 (2.35) | -0.2 (2.38)
  Maximum post BL, Sodium, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Sodium, n=888,866 | 0.6 (2.15) | 0.7 (2.22)
  Week 24, Urea, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Urea, n=839,787 | 0.08 (1.591) | 0.04 (1.549)
  Maximum post BL, Urea, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Urea, n=888,866 | 0.68 (1.601) | 0.64 (1.604)

43. Secondary Outcome: Change From Baseline in Glucose, Calcium, CO2, Chloride, Magnesium, Phosphate, Potassium, Sodium, and Urea at Week 52
Description: Blood samples were collected for the measurement of Glucose, calcium, CO2, chloride, magnesium, phophate, potassium, sodium, and urea at Baseline, Week 12, Week 24, and Week 52 for the extension part of the study. Change from Baseline was calculated as the post-Baseline value at Week 52 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: Mmol/L
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Mmol/L
  Week 52, Calcium, n=180,174: number analyzed (Participants) | 180 | 174
  Week 52, Calcium, n=180,174 | -0.033 (0.0943) | -0.040 (0.0968)
  Maximum post BL,Calcium, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Calcium, n=207,214 | 0.026 (0.0849) | 0.008 (0.0868)
  Week 52, Chloride, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Chloride, n=181,174 | -0.1 (3.00) | -0.2 (2.71)
  Maximum post BL,Chloride, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Chloride, n=207,214 | 1.4 (2.63) | 1.3 (2.39)
  Week 52, CO2, n=180,174: number analyzed (Participants) | 180 | 174
  Week 52, CO2, n=180,174 | -1.2 (2.46) | -1.0 (2.58)
  Maximum post BL,CO2, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,CO2, n=207,214 | -0.2 (2.26) | 0.3 (2.28)
  Week 52, Glucose, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Glucose, n=181,174 | 0.31 (1.538) | 0.22 (1.546)
  Maximum post BL,Glucose, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Glucose, n=207,214 | 0.92 (1.683) | 0.63 (1.738)
  Week 52, Potassium, n=180,174: number analyzed (Participants) | 180 | 174
  Week 52, Potassium, n=180,174 | -0.02 (0.443) | -0.10 (0.454)
  Maximum post BL,Potassium, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Potassium, n=207,214 | 0.29 (0.456) | 0.20 (0.418)
  Week 52, Phosphate, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Phosphate, n=181,174 | -0.003 (0.1645) | 0.005 (0.1800)
  Maximum post BL,Phosphate, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Phosphate, n=207,214 | 0.109 (0.1551) | 0.110 (0.1770)
  Week 52, Sodium, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Sodium, n=181,174 | -0.2 (2.34) | -0.1 (2.51)
  Maximum post BL,Sodium, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL,Sodium, n=207,214 | 1.1 (2.13) | 1.1 (2.22)
  Week 52, Urea, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Urea, n=181,174 | 0.16 (1.625) | 0.12 (1.553)
  Maximum post BL, Urea, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Urea, n=207,214 | 1.06 (1.755) | 1.08 (1.629)

44. Secondary Outcome: Change From Baseline in Bilirubin, Creatinine, and Urate at Week 24
Description: Blood samples were collected for the measurement of bilirubin, creatinine, and urate at Baseline, Week 12, and Week 24. Change from Baseline was calculated as the post-Baseline value at Week 24 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat). Only participants with data available at the analysis time point were analyzed (represented as n=X, X in category title). The maximum post-Baseline values have also been presented.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Micromoles per liter
  Week 24, Bilirubin, n=839,786: number analyzed (Participants) | 839 | 786
  Week 24, Bilirubin, n=839,786 | -0.2 (3.88) | 0.1 (3.77)
  Maximum post BL, Bilirubin, n=888,865: number analyzed (Participants) | 888 | 865
  Maximum post BL, Bilirubin, n=888,865 | 1.1 (4.09) | 1.2 (3.67)
  Week 24, Creatinine, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Creatinine, n=839,787 | 1.05 (9.816) | 1.14 (9.580)
  Maximum post BL, Creatinine, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Creatinine, n=888,866 | 4.12 (9.711) | 3.99 (9.509)
  Week 24, Urate, n=839,787: number analyzed (Participants) | 839 | 787
  Week 24, Urate, n=839,787 | 2.8 (60.87) | 1.7 (62.96)
  Maximum post BL, Urate, n=888,866: number analyzed (Participants) | 888 | 866
  Maximum post BL, Urate, n=888,866 | 23.7 (58.64) | 21.9 (59.20)

45. Secondary Outcome: Change From Baseline in Bilirubin, Creatinine, and Urate at Week 52
Description: Blood samples were collected for the measurement of bilirubin, creatinine, and urate at Baseline, Week 12, Week 24, and Week 52 of the extension part of the study. Change from Baseline was calculated as the post-Baseline value at Week 52 minus the Baseline value. Baseline was defined as the most recent individual value prior to randomization (generally Screening but could be a test repeat).
Time Frame: Baseline and Week 52
Population: Extension Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Micromoles per liter
  Week 52, Bilirubin, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Bilirubin, n=181,174 | 0.3 (3.41) | 0.1 (3.94)
  Maximum post BL, Bilirubin, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Bilirubin, n=207,214 | 2.0 (3.88) | 2.3 (4.28)
  Week 52, Creatinine, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Creatinine, n=181,174 | 2.95 (11.663) | 1.28 (11.563)
  Maximum post BL, Creatinine, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Creatinine, n=207,214 | 6.99 (11.425) | 6.00 (11.392)
  Week 52, Urate, n=181,174: number analyzed (Participants) | 181 | 174
  Week 52, Urate, n=181,174 | 3.6 (60.92) | 3.9 (64.85)
  Maximum post BL, Urate, n=207,214: number analyzed (Participants) | 207 | 214
  Maximum post BL, Urate, n=207,214 | 42.0 (62.06) | 40.0 (63.47)

46. Secondary Outcome: Number of Participants Reporting an Adverse Event of Special Interest (AESI) of Oropharyngeal Origin in the Treatment Period
Description: Oropharyngeal examinations for clinical evidence of infection (e.g., Candida albicans) were performed at each clinic visit. All suspected cases of candidiasis were reported as AEs. The number of participants with oral candidiasis, Candida infection, oral fungal infection, and oropharyngeal candidiasis were reported.
Time Frame: Up to Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Participants
  Oral candidiasis | 2 | 4
  Candida infection | 1 | 4
  Oral fungal infection | 2 | 3
  Oropharyngeal candidiasis | 2 | 0

47. Secondary Outcome: Number of Participants Reporting an AESI of Oropharyngeal Origin in the Extension Part of the Study
Description: as for outcome 46
Time Frame: Up to Week 52
Population: Extension Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Participants
  Candida infection | 0 | 3
  Oral fungal infection | 0 | 2

48. Secondary Outcome: Number of Participants With at Least One On-treatment Bone Fracture Incident in the Treatment Period
Description: To evaluate the potential for bone systemic corticosteroid effects, the incidence of bone fractures was assessed. It was categorized as an adverse event of special interest.
Time Frame: Up to Week 24
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 911 | 899
Participants | 4 | 6

49. Secondary Outcome: Number of Participants With at Least One On-treatment Bone Fracture Incident in the Extension Part of the Study
Description: as for outcome 48
Time Frame: Up to Week 52
Population: Extension Population
Measure: Number; unit: Participants
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Number analyzed (Participants) | 210 | 220
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from start of the study drug until Week 24 and follow-up period for participants in ITT population and up to Week 52 and follow-up for participants in Extension Population
Description: On-treatment SAEs and non-serious AEs are reported for ITT and extension populations
Arm/Group | FF/UMEC/VI 100/62.5/25 µg | BUD/FOR 400/12 µg
Serious Adverse Events (participants affected / at risk) | 61/911 | 64/899
Other Adverse Events (participants affected / at risk) | 105/911 | 104/899
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 µg (N=911) | BUD/FOR 400/12 µg (N=899)
Acute coronory syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Myocaridal ischemia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Catheter site phlebitis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Infective exacerbation of chronic onstructive airways diseas (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Intervertebra; disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brian neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischemic stroke (Nervous system disorders) | 1 | 0
Postical paralysis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Transient ischemic stroke (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Chronic kideny disease (Renal and urinary disorders) | 0 | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 31
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Heart valve replacement (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/UMEC/VI 100/62.5/25 µg (N=911) | BUD/FOR 400/12 µg (N=899)
Nasopharyngitis (Infections and infestations) | 72 | 51
Headache (Nervous system disorders) | 44 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.